CLINICAL TRIAL: NCT05604794
Title: Retrospective Review of Ketamine Assisted Psychotherapy Program on Mental Health at Field Trip Health Centres in North America
Brief Title: A Retrospective Effectiveness Trial of Ketamine-Assisted Psychotherapy in Adult Patients Coping With Mental Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Field Trip Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-3067-11240-5
Record Dates: First submitted 2022-10-12; First posted 2022-11-03 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Depression; Anxiety; Post Traumatic Stress Disorder
Keywords: ketamine; psychotherapy; mental health
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clients (Experimental): Adult patients coping with symptoms of depression, anxiety, and post traumatic stress
  Interventions: Combination Product: Ketamine-Assisted Psychotherapy (KAP)

INTERVENTIONS:
Combination Product: Ketamine-Assisted Psychotherapy (KAP) — KAP consisting of 4-6 guided ketamine sessions with psychotherapy-only visits after dose 1 and 2 and then after every 2 subsequent doses.

SUMMARY:
Ketamine-Assisted Psychotherapy (KAP) is a relatively new approach for the treatment of mental health issues, which involves the combination of ketamine, a dissociative anaesthetic with psychedelic properties, and psychotherapy to promote emotional wellbeing. In this study, we investigated the effectiveness of KAP in adult patients coping with mental health. We predicted that clients would experience lasting reductions in psychological distress over time, such as depression, anxiety, and post traumatic stress, that would be detectable up to 6 months after treatment. The results of this study may provide evidence of sustained real-world effects of Ketamine-Assisted Psychotherapy, of interest to patients, clinicians, researchers, and policymakers.

DETAILED DESCRIPTION:
Background: Ketamine-Assisted Psychotherapy (KAP) has shown positive effects within clinical trial settings and over short-term follow-ups, but sustained effects in real-world treatment settings remain unclear. In this study, we investigated the effectiveness of KAP in adult patients coping with mental health issues. We hypothesized that there would be significant reductions in psychological distress over time.

Objective: To examine treatment effects at 1, 3, and 6 months relative to baseline on depression, anxiety, and post traumatic stress outcomes.

Design: A retrospective intervention-only effectiveness trial.

Setting: KAP was administered across 11 Field Trip Health clinics in North America. Intervention: KAP consisting of 4-6 guided ketamine sessions with psychotherapy-only visits after dose 1 and 2 and then after every 2 subsequent doses.

Outcomes: Self-reported measures of symptoms of depression, anxiety, and post traumatic stress at 1, 3, and 6 months.

Statistical Analysis: Analyses were by intention to treat. Main analysis was a mixed linear model or growth curve model to estimate change over time per outcome, yielding estimates of mean changes at each endpoint relative to baseline. Secondary analyses included evaluating case reductions (identified by cut-off values) and minimal clinically important differences (MCIDs) at each endpoint relative to baseline.

Significance: This study may provide evidence of sustained real-world effects of Ketamine-Assisted Psychotherapy, of interest to patients, clinicians, researchers, and policymakers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Over the age of 18
* Should be psychologically and medically cleared by a psychiatrist, family physician, or treatment team
* Diagnosed with Major Depressive Disorder (MDD), Bipolar Depression, Generalized Anxiety Disorder, Obsessive Compulsive Disorder (OCD), and Eating Disorder by a licensed healthcare practitioner (including Field Trip Consultants)
* A significant history of trauma and/or formal diagnosis of PTSD as per the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5)
* Individuals who have received Electroconvulsive Therapy (ECT) or other neuromodulatory treatments like Transcranial Magnetic Stimulation (TMS)
* Individuals reporting suicidal ideation may be included, as suicidal ideation is a symptom of a Major Depressive Episode (MDE)

Exclusion Criteria:

* Individuals who are unable to consent to the treatment
* Pregnant women and nursing mothers

  --Note that Post Partum Depression (PPD) can be considered on a case-by-case basis in consultation with the National Medical Director.
* There is a relative (not absolute) contraindication for individuals with a Body Mass Index (BMI) of above 35. These clients must be given thorough consideration by the medical team.
* Any individual who has met DSM 5 criteria for a Substance Use Disorder in the past 3 months.

  * Note that patients with alcohol, opioid, benzodiazepine, cocaine, and amphetamine use disorders need to go through detox (for alcohol/benzodiazepines) and be sober for 4 weeks.
  * Note that mild active alcohol, cocaine, and cannabis use can be considered on a case-by-case basis at the comfort level of the treatment team if the client has demonstrated abstaining or significant reduction of use prior to starting treatment.
* Daily use of moderate to high doses of benzodiazepines
* Individuals who are experiencing psychotic symptoms as part of an MDE (mood congruent/ mood incongruent)
* Psychosis: Schizophrenia, Schizoaffective disorder, Bipolar 1 with psychotic features during mania
* Active Mania: Bipolar 1 (chronic non-disruptive hypomania is an exception at the discretion of the consultant)
* Borderline Personality Disorder
* Uncontrolled medical disorders
* Physical conditions with negative interaction with ketamine (e.g., metabolic blood disorder)
* Individuals with symptomatic acute brain injury within 90 days of serious injury
* Individuals diagnosed with moderate to severe sleep apnea
* Individuals who are unable to identify a person or service to assure their safe transport to home post treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1806 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Yermus, MD, Principal Investigator — Field Trip Health; Chris Lo, PhD, Principal Investigator — University of Toronto
Locations (11):
- United States (8):
  - LA Centre, Los Angeles, California
  - San Diego Centre, San Diego, California
  - Washington DC Centre, Washington D.C., District of Columbia
  - Atlanta Centre, Atlanta, Georgia
  - Chicago Centre, Chicago, Illinois
  - NYC Centre, New York, New York
  - Houston Centre, Houston, Texas
  - Seattle Centre, Seattle, Washington
- Canada (3):
  - Vancouver Centre, Vancouver, British Columbia
  - Fredericton Centre, Fredericton, New Brunswick
  - Field Trip Health, Toronto Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clients
Started | 1806
Completed | 94
Not Completed | 1712

BASELINE CHARACTERISTICS:
Arm/Group | Clients
Number analyzed (Participants) | 1806
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 948
  Gender: Male | 850
  Gender: Non-binary | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 1309
  Race/Ethnicity: Other Groups | 441
  Race/Ethnicity: Missing | 56
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 1806

OUTCOME MEASURES:

1. Primary Outcome: 9-item Patient Health Questionnaire (PHQ-9)
Description: Self-reported measure of depression, ranging from 0-27. Higher scores are worse.
Time Frame: Change from 3 months compared to baseline
Population: Number analysed after attrition.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 315
units on a scale | -3.23 [-3.57 to -2.90]

2. Primary Outcome: 7-item Generalized Anxiety Disorder Measure (GAD-7)
Description: Self-reported measure of anxiety, ranging from 0-21. Higher scores are worse.
Time Frame: Change from 3 months compared to baseline
Population: Number analysed after attrition.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 305
units on a scale | -4.80 [-5.17 to -4.44]

3. Primary Outcome: 6-item PTSD Checklist (PCL-6)
Description: Self-reported measure of post traumatic stress, ranging from 6-30. Higher scores are worse.
Time Frame: Change from 3 months compared to baseline
Population: Number analysed after attrition.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 299
units on a scale | -4.24 [-4.60 to -3.87]

4. Secondary Outcome: 9-item Patient Health Questionnaire (PHQ-9)
Description: Self-reported measure of depression, ranging from 0-27.
Time Frame: Change from 1 month compared to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 330
units on a scale | -3.23 [-3.57 to -2.90]

5. Secondary Outcome: 9-item Patient Health Questionnaire (PHQ-9)
Description: Self-reported measure of depression, ranging from 0-27.
Time Frame: Change from 6 months compared to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 92
units on a scale | -4.74 [-5.68 to -3.80]

6. Secondary Outcome: 7-item Generalized Anxiety Disorder Measure (GAD-7)
Description: Self-reported measure of anxiety, ranging from 0-21.
Time Frame: Change from 1 month compared to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 333
units on a scale | -2.65 [-2.95 to -2.34]

7. Secondary Outcome: 7-item Generalized Anxiety Disorder Measure (GAD-7)
Description: Self-reported measure of anxiety, ranging from 0-21.
Time Frame: Change from 6 months compared to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 72
units on a scale | -4.10 [-5.02 to -3.18]

8. Secondary Outcome: 6-item PTSD Checklist (PCL-6)
Description: Self-reported measure of post traumatic stress, ranging from 6-30.
Time Frame: Change from 1 month compared to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 327
units on a scale | -2.14 [-2.44 to -1.83]

9. Secondary Outcome: 6-item PTSD Checklist (PCL-6)
Description: Self-reported measure of post traumatic stress, ranging from 6-30.
Time Frame: Change from 6 months compared to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Clients
Number analyzed (Participants) | 69
units on a scale | -3.44 [-4.38 to -2.50]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Clients
All-Cause Mortality (participants affected / at risk) | 0/1806
Serious Adverse Events (participants affected / at risk) | 0/1806
Other Adverse Events (participants affected / at risk) | 0/1806

LIMITATIONS AND CAVEATS:
Based on feedback from the peer review process, this study should be considered a cohort study rather than a trial. The high attrition rate may limit validity of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT05604794/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT05604794/ICF_000.pdf